CLINICAL TRIAL: NCT03419637
Title: Evaluating the Use of Mobile Devices as Educational Tools Regarding Skin History
Brief Title: Mobile Devices as Educational Skin History Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 826558
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard of Care (No Intervention): The standard of care consists of in-clinic counseling, informational handouts, and access to patient medical records
- Intervention - Mobile app (Experimental): The mobile app, or app, is used to document before and after photos of the excised skin areas and to document related diagnoses. The app allows patients to view a skin history summary report and a reference on their skin ﬁndings and procedures.
  Interventions: Other: Mobile app

INTERVENTIONS:
Other: Mobile app — The mobile app, or app, is installed on the patient's mobile device and is used to document the surgical procedure with before and after photographs, including pre- and post-surgery diagnosis. The app allows patients to view a skin history summary report and a reference on their skin ﬁndings and procedures.
  Arms: Intervention - Mobile app

SUMMARY:
Part I of this study surveys patients in the Penn Dermatologic Surgery Clinic to evaluate if a need exists for increased patient understanding of their skin history and which factors, if any, related to the patient or their skin history are associated with this need. In part II, the study aim is to evaluate mobile technology as a way of improving patient understanding of diagnoses, treatments, and procedures. In this part of the study, eligible patients from part I will be randomized either to a control group that receives the current standard of care regarding in-clinic counseling, informational handouts, and access to their medical records, or to an intervention group that in addition to the current standard of care, is setup with a mobile app, allowing patients to view a skin history summary report and a reference on their skin ﬁndings and procedures. Patients then complete a survey to establish their baseline understanding of their clinic visit. Three weeks later the patient is emailed a follow-up survey to assess their understanding of their in-clinic visit. Differences in understanding between the two study groups will be assessed by comparing the number of correctly answered survey items regarding their in-clinic visit, both at baseline (immediately following their surgery) and three weeks later. Qualitative information regarding satisfaction and areas of improvement will also be collected via survey. Patients who have an appointment during the study period at the Penn Dermatologic Surgery clinic for a skin excision will be eligible for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Have an appointment in the Penn Dermatologic Surgery Clinic for removal of a skin area during the study enrollment period
* Possession of a mobile device running iOS with the study mobile app (intervention) successfully installed (assistance will be provided by research staff if needed)

Exclusion Criteria:

* Children or adolescents, or if the patient is court-ordered to attend residential alcohol or other drug treatment facilities and therefore considered prisoners
* Patients will also be excluded if they are incompetent to provide informed consent and HIPAA authorization.
* If the area being operated on is of the genitals or breasts
* If the area being operated on is of the face, and photos of the area cannot be cropped or the eyes cannot be covered sufﬁciently such that photos are non-identifying

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Understanding of recent skin excision - 3 weeks later | 3 weeks
  After study enrollment, patients have one or more skin areas excised. They complete an in-clinic survey immediately after the excision and another survey 3 weeks later where they are asked questions regarding the clinic visit and the related excised skin areas and diagnoses. Understanding is assessed by comparing against the medical record to calculate the number/percent of correct responses.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Miller, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No